CLINICAL TRIAL: NCT04301245
Title: Profile of COPD Patients Refusing Educational Program in Pulmonary Rehabilitation and Impact on the Benefits
Status: Completed | Type: Observational
Sponsor: ADIR Association (Other)
Responsible Party: Sponsor
Other Study IDs: RETRO-ETP
Record Dates: First submitted 2020-03-06; First posted 2020-03-10 (Actual); Last update posted 2020-06-01 (Actual); Status verified 2020-05

CONDITIONS: Chronic Obstructive Pulmonary Disease; Pulmonary Rehabilitation
Keywords: Chronic Obstructive Pulmonary Disease; Pulmonary Rehabilitation; Education
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ETEP group: Exercise Training and Educational Program (ETEP) group. Patients who accepted the educational program in addition to the exercise training.
  Interventions: Other: Educational program
- ET group: Exercise Training (ET) group. Patients who refused the educational program and did only the exercise training.
  Interventions: Other: Educational program

INTERVENTIONS:
Other: Educational program — The educational program (EP) was offered during the initial session of the pulmonary rehabilitation. According to the french law, patients were free to participate or not.
  The EP consisted of an educational diagnosis, educational workshops and an individual final assessment.

SUMMARY:
Pulmonary rehabilitation (PR) has proven its efficacy to improve dyspnea, health status, exercise tolerance and quality of life for patients with stable Chronic Obstructive Pulmonary Disease (COPD). Exercise training has previously been thoroughly studied but education has been less studied in PR. Furthermore, only few studies have investigated the added value of an educational program (EP) to exercise training on clinical and physical factors. Characterizing those patients who refuse EP is therefore a first step to better target them and potentially improve their adherence and outcome following PR.

The aim of this study was to determine the characteristics of the COPD patients referred to PR who refused EP compare to those who accepted and to identify the independent predictive factors of refusal. The investigators also sought to compare the change in clinical outcomes and number and length of hospitalization at six months following PR among those patients who accepted or not to participate in EP.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of COPD,
* >18 years old,
* Stable state of COPD.

Exclusion Criteria:

* Patients who have not been offered an educational program
* Patients who have already been offered an educational program during a pulmonary rehabilitation in the same center.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred for pulmonary rehabilitation between July 2015 and July 2019 to ADIR Association, Rouen University Hospital, France
Sampling Method: Non-Probability Sample
Enrollment: 201 (Actual)
Dates: Start 2020-02-28 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-04-10 (Actual)

PRIMARY OUTCOMES:
Multiple logistic regression between the variables defined and the refusal of educational program | Baseline
  The variables are described below in primary outcomes
Gender | Baseline
  Gender will be analysed in logistic regression.
Age | Baseline
  Age will be analysed in logistic regression.
Height | Baseline
  Height will be analysed in logistic regression.
Weight | Baseline
  Weight will be analysed in logistic regression.
Body mass index | Baseline
  Body mass index will be analysed in logistic regression.
COPD stages | Baseline
  COPD stages will be analysed in logistic regression.
Forced Expiratory Volume in one second | Baseline
  Forced Expiratory Volume in one second will be analysed in logistic regression.
Forced Vital Capacity | Baseline
  Forced Vital Capacity will be analysed in logistic regression.
Ratio between Forced Expiratory Volume in one second and Forced Vital Capacity | Baseline
  Ratio between Forced Expiratory Volume in one second and Forced Vital Capacity will be analysed in logistic regression.
Total Lung Capacity | Baseline
  Total Lung Capacity will be analysed in logistic regression.
Residual Volume | Baseline
  Residual Volume will be analysed in logistic regression.
Diffusing capacity of the lungs for carbon monoxide divided by alveolar volume | Baseline
  Diffusing capacity of the lungs for carbon monoxide divided by alveolar volume will be analysed in logistic regression.
Comorbidities | Baseline
  Comorbidities will be analysed in logistic regression.
Tabacco status | Baseline
  Tabacco status will be analysed in logistic regression.
Tabacco consumption | Baseline
  Tabacco consumption will be analysed in logistic regression.
Prescription of oxygen | Baseline
  Prescription of oxygen will be analysed in logistic regression.
Prescription of non invasive ventilation | Baseline
  Prescription of non invasive ventilation will be analysed in logistic regression.
Arterial oxygen partial pressure | Baseline
  Arterial oxygen partial pressure will be analysed in logistic regression.
Arterial carbon dioxide partial pressure | Baseline
  Arterial carbone dioxide partial pressure will be analysed in logistic regression.
Location of the training sessions | Baseline
  Location of the training sessions will be analysed in logistic regression.
Ambulance transport | Baseline
  Number of patients with an ambulance transport will be analysed in logistic regression.
Distance between patient's home and center | Baseline
  Distance between patient's home and center will be analysed in logistic regression.
Dyspnea | Baseline
  Dyspnea assessed by the modified Medical Research Council scale will be analysed in logistic regression.
6-Minute Stepper Test | Baseline
  Number of steps during the 6-Minute Stepper Test will be analysed in logistic regression.
6-Minute Walk Test | Baseline
  Distance during the 6-Minute Walk Test will be analysed in logistic regression.
Maximal oxygen consumption | Baseline
  Maximal oxygen consumption during cardiopulmonary exercise testing will be analysed in logistic regression.
Maximal workload | Baseline
  Maximal workload achieved during cardiopulmonary exercise testing will be analysed in logistic regression.
Saint George's Respiratory Questionnaire | Baseline
  Quality of life assessed by Saint George's Respiratory Questionnaire will be analysed in logistic regression.
Employment | Baseline
  Employment will be analysed in logistic regression.
Educational level | Baseline
  Educational level assessed by the international classification "Classification Internationale Type de l'Education" will be analysed in logistic regression.
Cognitive impairment | Baseline
  Cognitive impairment assessed by the Montreal Cognitive Assessment will be analysed in logistic regression.
Anxiety and depression level | Baseline
  Anxiety and depression level assessed by the Hospital Anxiety and Depression scale will be analysed in logistic regression.

SECONDARY OUTCOMES:
6-Minute Stepper Test | 2 months
  Change in number of steps during the 6-Minute Stepper Test will be compared between groups.
6-Minute Walk Test | 2 months
  Change in distance during the 6-Minute Walk Test will be compared between groups.
Saint George's Respiratory Questionnaire | 2 months
  Change in Saint George's Respiratory Questionnaire will be compared between groups.
Anxiety and depression level | 2 months
  Anxiety and depression level assessed by the Hospital Anxiety and Depression scale will be analysed in logistic regression.
Cognitive impairment | 2 months
  Change in cognitive impairment assessed by the Montreal Cognitive Assessment will be compared between groups.
Number of hospitalizations | 6 months
  Number of hospitalizations will be compared between groups.
Number of hospitalized patients | 6 months
  Number of hospitalized patients will be compared between groups.
Number of days of hospitalization | 6 months
  Number of days of hospitalization will be compared between groups.
Attendance rate at educational sessions | 2 months
  Attendance rate at education sessions will be analysed

CONTACTS AND LOCATIONS:
Overall Officials: Jean-François Muir, MD PhD, Principal Investigator — ADIR Association, Rouen University Hospital, Rouen, France;Normandie University, UNIROUEN, UPRES EA 3830, Rouen University Hospital, Haute-Normandie Research and Biomedical Innovation, Rouen, France; Antoine Cuvelier, MD PhD, Study Chair — Normandie University, Rouen University Hospital, Haute-Normandie Research and Biomedical Innovation, Rouen, France ; Pulmonary, Thoracic Oncology and Respiratory Intensive Care Department, Rouen University Hospital, Rouen, France.; David Debeaumont, MD, Study Chair — Department of Respiratory and Exercise Physiology and CICCRB 1404, Rouen University Hospital, Rouen France.; Tristan Bonnevie, PT MSc, Study Chair — ADIR Association, Rouen University Hospital, Rouen, France ; Normandie University, UNIROUEN, UPRES EA 3830, Rouen University Hospital, Haute- Normandie Research and Biomedical Innovation, Rouen, France.; Francis-Edouard Gravier, PT MSc, Study Chair — ADIR Association, Rouen University Hospital, Rouen, France ; Normandie University, UNIROUEN, UPRES EA 3830, Rouen University Hospital, Haute- Normandie Research and Biomedical Innovation, Rouen, France; Pauline Smondack, PT, Study Chair — ADIR Association, Rouen University Hospital, Rouen, France.
Locations (1):
- ADIR Association, Bois-Guillaume, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Smondack P, Gravier FE, Combret Y, Muir JF, Cuvelier A, Debeaumont D, Medrinal C, Prieur G, Bonnevie T. Factors influencing participation in educational workshops as part of a pulmonary rehabilitation program in patients with chronic obstructive pulmonary disease: a retrospective study. Expert Rev Respir Med. 2022 Mar;16(3):341-349. doi: 10.1080/17476348.2022.1991793. Epub 2021 Nov 2. PMID 34623218